CLINICAL TRIAL: NCT00951015
Title: A Phase IIb Study to Select a Once Daily Dose of GSK1349572 Administered With Either Abacavir/Lamivudine or Tenofovir/Emtricitabine in HIV-1 Infected Antiretroviral Therapy Naive Adult Subjects
Brief Title: A Dose Ranging Trial of GSK1349572 and 2 NRTI in HIV-1 Infected, Therapy Naive Subjects
Acronym: ING112276
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112276
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-04

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1349572; emtricitabine; tenofovir; efavirenz; abacavir; antiretroviral therapy naive; dose selection; HIV-1 Infection; integrase inhibitor; HIV infection; once daily; lamivudine
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mg GSK1349572 (Experimental): subjects will receive GSK1349572 10mg once daily blinded to dose
  Interventions: Drug: GSK1349572
- 25mg GSK1349572 (Experimental): subjects will receive GSK1349572 25mg once daily blinded to dose
  Interventions: Drug: GSK1349572
- 50mg GSK1349572 (Experimental): subjects will receive GSK1349572 50mg once daily blinded to dose
  Interventions: Drug: GSK1349572
- efavirenz control (Other): efavirenz will serve as the internal control arm
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: GSK1349572 — investigational HIV-1 integrase inhibitor
  Arms: 10 mg GSK1349572; 25mg GSK1349572; 50mg GSK1349572
Drug: efavirenz — approved therapy for HIV-1 infection, used as an internal study control
  Arms: efavirenz control

SUMMARY:
This Phase IIb study in HIV-infected antiretroviral naive subjects will select an optimal once daily dose of GSK1349572 from a range of doses for future evaluation.

DETAILED DESCRIPTION:
This Phase IIb study in HIV-infected antiretroviral naive adult subjects will include a dose-ranging evaluation of GSK1349572 10mg, 25mg and 50mg once daily blinded doses and a control arm of open label efavirenz 600mg once daily. Background ART for all study subjects will be chosen by the investigators and will be either Truvada or Epzicom/Kivexa. Data from the three doses of GSK1349572 will be compared on the basis of antiviral activity, safety/tolerability and pharmacokinetics over 16-24 weeks.

Several planned interim analyses will evaluate data in real time; any doses considered inferior will be dropped and subjects on those doses of GSK1349572 will have the option to switch to either the highest dose still under investigation or the selected dose. Subjects will be able to remain in the study, unless they reach a stopping criterion, for at least 96 weeks.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected male or female adults at least 18 years of age. Women capable of becoming pregnant must use appropriate contraception during the study (as defined by the protocol);
* HIV-1 infection with a screening plasma HIV-1 RNA greater than or equal to 1000copies/mL;
* CD4+ cell count greater than or equal to 200cells/mm3 (or higher as local guidelines dictate);
* ART-naive (less than or equal to 10 days of prior therapy with any antiretroviral agent). Any previous exposure to an HIV integrase inhibitor other than GSK1349572 will be exclusionary.
* No evidence of viral resistance to any antiretroviral drug indicative of primary transmitted resistance at screening;
* Able to understand and comply with protocol requirements;
* Able to provide written informed consent prior to screening;
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Note: Subjects starting abacavir as part of the NRTI backbone must have been screened and be negative for the HLA-B*5701 allele.

Exclusion Criteria:

* Any pre-existing or serious mental or physical disorder which could compromise ability to comply with the protocol or compromise subject safety;
* Women who are pregnant or breastfeeding;
* An active AIDS-defining condition at the screening visit;
* Previous participation in an experimental drug and/or vaccine trial(s) within 30 days or 5 half-lives;
* History of clinically relevant pancreatitis or hepatitis within the previous 6 months, including HBsAg positive result. Asymptomatic HCV infection will not be exclusionary, however subject who will require HCV therapy during the trial should be excluded. Any subject with a history of liver cirrhosis with or without hepatitis viral co-infection will be excluded.
* Any condition which could interfere with the absorption, distribution, metabolism or excretion of the drug;
* Any acute or Grade 4 laboratory abnormality at screening;
* History of upper gastrointestinal bleed and/or subjects with active peptic ulcer disease;
* Estimated creatinine clearance <50 mL/min;
* Alanine aminotransferase (ALT) greater than or equal to 5 times ULN;
* Alanine aminotransferase (ALT) greater than or equal to 3xULN and bilirubin greater than or equal to 1.5xULN (with >35% direct bilirubin);
* Lipase greater than or equal to 3xULN;
* Hemoglobin < 100 g/L(10 g/dL);
* History of allergy to the study drugs or their components or drugs of their class;
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents, any agents with activity against HIV-1 or immunomodulators within 28 days prior to screening;
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days prior to screening;
* History of protocol-defined cardiac diseases;
* Personal or family history of prolonged QT syndrome;
* Any clinically significant finding, as specified in the protocol, on electrocardiograph (ECG);
* Significant blood loss in excess of 500 mL within a 56 day period prior to screening visit;
* Immunization within 30 days prior to first dose of investigational product;
* French subjects: The subject has participated in any study using an investigational drug during the previous 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine - whichever is longer, prior to screening for the study or the subject will participate simultaneously in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-07-30; Primary Completion 2010-02-26 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (26):
- United States (11):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Dallas, Texas
- France (4):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hamburg
- Italy (3):
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
- Russia (2):
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- Spain (3):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

REFERENCES:
- [Background] van Lunzen J, Maggiolo F, Arribas JR, Rakhmanova A, Yeni P, Young B, Rockstroh JK, Almond S, Song I, Brothers C, Min S. Once daily dolutegravir (S/GSK1349572) in combination therapy in antiretroviral-naive adults with HIV: planned interim 48 week results from SPRING-1, a dose-ranging, randomised, phase 2b trial. Lancet Infect Dis. 2012 Feb;12(2):111-8. doi: 10.1016/S1473-3099(11)70290-0. Epub 2011 Oct 20. PMID 22018760

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization Phase participants received Dolutegravir (DTG 10, 25 or 50 milligrams[mg]) with Placebo/Efavirenz (EFV) for 96 Weeks . DTG participants who completed 96 Weeks continued or were switched to receive DTG 50 mg in Open label phase until DTG was locally available.
Pre-assignment Details: A total of 278 par were screened of which 70 were screen failures and 208 were randomized; 205 received at least one dose of study medication and comprised the Intent-To-Treat exposed (ITT-E) population. 17 participants out of 155 from DTG arm withdrew during Randomization phase and total 138 participants were enrolled in an Open-label phase.
Groups:
- DTG 10 mg QD: Participants received DTG 10 mg, DTG matching placebo, and Abacavir/lamivudine (ABC/3TC) 600 mg/300 mg or tenofovir/emtricitabine (TDF/FTC) 300 mg/200 mg orally once daily (QD) for 96 weeks.
- DTG 25 mg QD: Participants received DTG 25 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- DTG 50 mg QD: Participants received DTG 50 mg matching placebo and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- EFV 600 mg QD: Participants received Efavirenz (EFV) 600 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- Open-label DTG 50 mg QD: All DTG participants were switched to or continued DTG 50 mg with either ABC/3TC orally at 600 mg/300 mg (1 tablet) or TDF/FTC orally QD during the Open label phase
Period: Randomization Phase 96 Week
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD | Open-label DTG 50 mg QD
Started | 53 | 51 | 51 | 50 | 0
Completed | 48 | 44 | 46 | 40 | 0
Not Completed | 5 | 7 | 5 | 10 | 0
Not completed — Adverse Event | 1 | 1 | 2 | 5 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 0
Not completed — Protocol-Defined Stopping Criteria | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 3 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2 | 0
Period: Open-label Phase
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD | Open-label DTG 50 mg QD
Started | 0 | 0 | 0 | 0 | 138
Completed | 0 | 0 | 0 | 0 | 88
Not Completed | 0 | 0 | 0 | 0 | 50
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 12
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 14
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- DTG 10 mg QD: Participants received Dolutegravir (DTG) 10 milligrams (mg), DTG matching placebo, and Abacavir (ABC)/Lamivudine (3TC) 600 mg/300 mg or Tenofovir (TDF)/Emtricitabine (FTC) 300 mg/200 mg orally once daily (QD) for 96 weeks.
- DTG 50 mg QD: Participants received DTG 50 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- Total: Total of all reporting groups
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD | Total
Number analyzed (Participants) | 53 | 51 | 51 | 50 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (9.25) | 37.0 (9.79) | 37.0 (8.89) | 40.7 (11.19) | 37.2 (10.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 6 | 6 | 28
  Male | 42 | 46 | 45 | 44 | 177
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage (HER) | 7 | 6 | 8 | 4 | 25
  American Indian or Alaska Native | 1 | 3 | 4 | 2 | 10
  Japanese/East Asian HER/South East Asian HER | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 3 | 0 | 0 | 0 | 3
  White | 41 | 42 | 38 | 43 | 164
  African American/African HER & White | 0 | 0 | 1 | 0 | 1
  Asian & White | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/Milliliter (c/mL) at Week 16
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Week 16. The analysis was performed using the time to loss of virological response (TLOVR) dataset. In the TLOVR dataset, participant responses at a specified threshold of HIV-1 RNA (<50 copies/mL) are determined by using the Food and Drug Administration's TLOVR algorithm. Using the TLOVR algorithm, participants are considered to have failed on therapy if they never achieved confirmed RNA levels below the threshold, if they had confirmed rebound of RNA above the threshold, if they made a non-permitted change in background regimen, or if they permanently discontinued investigational product for any reason. Data are reported per the Week 16 report. In later cuts of the data, the Week 16 values may have changed (because of the nature of the TLOVR algorithm).ITT-E Population included all randomized participants who received at least one dose of study medication
Time Frame: Week 16
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
participants | 51 | 47 | 46 | 29

2. Secondary Outcome: Viral Change Over the Initial 2 Weeks of Treatment
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline and Week 2. Viral change is defined as the change in plasma HIV-1 RNA over the initial 2 weeks of treatment, calculated as the value at Week 2 minus the value at Baseline. Only those participants available at the specified time point were analyzed.
Time Frame: Baseline and Week 2
Population: ITT-E Population.
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Groups:
- DTG 10 mg QD: Participants received DTG 10 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 50 | 50 | 48
Log10 c/mL | -2.387 (0.4595) | -2.365 (0.5458) | -2.392 (0.4241) | -1.930 (0.4312)

3. Secondary Outcome: Change From Baseline in HIV-1 RNA at the Indicated Time Points
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1), Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, Week 84, and Week 96. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline (Day 1), Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, Week 84, and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT-E Population.
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Log10 c/mL
  Week 1, n=53, 50, 48, 50: number analyzed (Participants) | 53 | 50 | 48 | 50
  Week 1, n=53, 50, 48, 50 | -1.815 (0.3999) | -1.773 (0.4650) | -1.738 (0.3840) | -1.562 (0.4158)
  Week 2, n=53, 50, 50, 48: number analyzed (Participants) | 53 | 50 | 50 | 48
  Week 2, n=53, 50, 50, 48 | -2.387 (0.4595) | -2.365 (0.5458) | -2.392 (0.4241) | -1.930 (0.4312)
  Week 4, n=53, 50, 50, 45: number analyzed (Participants) | 53 | 50 | 50 | 45
  Week 4, n=53, 50, 50, 45 | -2.629 (0.5863) | -2.583 (0.6337) | -2.713 (0.5471) | -2.162 (0.5400)
  Week 8, n=52, 50, 49, 45: number analyzed (Participants) | 52 | 50 | 49 | 45
  Week 8, n=52, 50, 49, 45 | -2.657 (0.6980) | -2.666 (0.6667) | -2.848 (0.6556) | -2.450 (0.5989)
  Week 12, n=53, 49, 49, 45: number analyzed (Participants) | 53 | 49 | 49 | 45
  Week 12, n=53, 49, 49, 45 | -2.685 (0.6831) | -2.671 (0.6850) | -2.860 (0.6772) | -2.603 (0.5869)
  Week 16, n=52, 49, 49, 45: number analyzed (Participants) | 52 | 49 | 49 | 45
  Week 16, n=52, 49, 49, 45 | -2.718 (0.6593) | -2.668 (0.6826) | -2.859 (0.6876) | -2.698 (0.6715)
  Week 20, n=52, 48, 49, 44: number analyzed (Participants) | 52 | 48 | 49 | 44
  Week 20, n=52, 48, 49, 44 | -2.701 (0.6423) | -2.662 (0.6908) | -2.869 (0.6896) | -2.745 (0.6602)
  Week 24, n=52, 49, 48, 45: number analyzed (Participants) | 52 | 49 | 48 | 45
  Week 24, n=52, 49, 48, 45 | -2.700 (0.6261) | -2.657 (0.6969) | -2.853 (0.6889) | -2.773 (0.7026)
  Week 32, n=52, 49, 47, 45: number analyzed (Participants) | 52 | 49 | 47 | 45
  Week 32, n=52, 49, 47, 45 | -2.717 (0.6588) | -2.658 (0.6991) | -2.855 (0.6963) | -2.772 (0.7021)
  Week 40, n=51, 48, 47, 44: number analyzed (Participants) | 51 | 48 | 47 | 44
  Week 40, n=51, 48, 47, 44 | -2.647 (0.7039) | -2.665 (0.7051) | -2.855 (0.6934) | -2.795 (0.7169)
  Week 48, n=51, 48, 48, 45: number analyzed (Participants) | 51 | 48 | 48 | 45
  Week 48, n=51, 48, 48, 45 | -2.723 (0.6519) | -2.667 (0.6934) | -2.850 (0.6849) | -2.711 (0.7765)
  Week 60, n=50, 48, 48, 44: number analyzed (Participants) | 50 | 48 | 48 | 44
  Week 60, n=50, 48, 48, 44 | -2.741 (0.6444) | -2.675 (0.7012) | -2.825 (0.7458) | -2.765 (0.7035)
  Week 72, n=51, 47, 48, 44: number analyzed (Participants) | 51 | 47 | 48 | 44
  Week 72, n=51, 47, 48, 44 | -2.742 (0.6453) | -2.622 (0.8052) | -2.860 (0.6930) | -2.757 (0.7094)
  Week 84, n=51, 47, 47, 43: number analyzed (Participants) | 51 | 47 | 47 | 43
  Week 84, n=51, 47, 47, 43 | -2.725 (0.6506) | -2.670 (0.7064) | -2.855 (0.6923) | -2.743 (0.7321)
  Week 96, n=48, 44, 46, 39: number analyzed (Participants) | 48 | 44 | 46 | 39
  Week 96, n=48, 44, 46, 39 | -2.728 (0.6494) | -2.680 (0.7116) | -2.854 (0.7061) | -2.807 (0.7238)

4. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Counts at the Indicated Time Points
Description: Blood samples were collected for lymphocyte subset assessment by flow cytometry at Baseline (Day 1), Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, Week 84, and Week 96. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT-E Population.
Time Frame: as for outcome 3
Population: ITT-E Population.
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Cells per cubic millimeter
  Week 1, n=53, 50, 48, 50: number analyzed (Participants) | 53 | 50 | 48 | 50
  Week 1, n=53, 50, 48, 50 | 85.0 [18.0 to 134.0] | 94.5 [40.0 to 160.0] | 75.5 [18.5 to 129.5] | 42.5 [-23.0 to 111.0]
  Week 2, n=53, 50, 50, 47: number analyzed (Participants) | 53 | 50 | 50 | 47
  Week 2, n=53, 50, 50, 47 | 75.0 [37.0 to 124.0] | 79.0 [27.0 to 138.0] | 99.5 [53.0 to 160.0] | 55.0 [-10.0 to 132.0]
  Week 4, n=53, 50, 50, 45: number analyzed (Participants) | 53 | 50 | 50 | 45
  Week 4, n=53, 50, 50, 45 | 75.0 [34.0 to 151.0] | 89.0 [36.0 to 165.0] | 110.0 [46.0 to 170.0] | 89.0 [30.0 to 165.0]
  Week 8, n=52, 50, 49, 44: number analyzed (Participants) | 52 | 50 | 49 | 44
  Week 8, n=52, 50, 49, 44 | 118.5 [65.5 to 210.5] | 156.5 [93.0 to 226.0] | 129.0 [105.0 to 201.0] | 104.5 [34.5 to 240.5]
  Week 12, n=53, 48, 48, 45: number analyzed (Participants) | 53 | 48 | 48 | 45
  Week 12, n=53, 48, 48, 45 | 139.0 [96.0 to 284.0] | 137.5 [61.0 to 250.0] | 171.5 [107.5 to 269.0] | 127.0 [58.0 to 186.0]
  Week 16, n=52, 49, 49, 44: number analyzed (Participants) | 52 | 49 | 49 | 44
  Week 16, n=52, 49, 49, 44 | 153.0 [95.0 to 276.0] | 176.0 [86.0 to 227.0] | 160.0 [94.0 to 227.0] | 115.5 [65.5 to 226.0]
  Week 20, n=52, 48, 49, 44: number analyzed (Participants) | 52 | 48 | 49 | 44
  Week 20, n=52, 48, 49, 44 | 163.5 [79.5 to 288.5] | 200.0 [103.0 to 316.5] | 139.0 [64.0 to 238.0] | 136.0 [54.5 to 215.5]
  Week 24, n=51, 49, 47, 44: number analyzed (Participants) | 51 | 49 | 47 | 44
  Week 24, n=51, 49, 47, 44 | 159.0 [97.0 to 233.0] | 206.0 [102.0 to 289.0] | 167.0 [125.0 to 268.0] | 109.5 [66.0 to 229.0]
  Week 32, n=50, 48, 47, 44: number analyzed (Participants) | 50 | 48 | 47 | 44
  Week 32, n=50, 48, 47, 44 | 221.5 [94.0 to 300.0] | 195.5 [109.0 to 294.0] | 203.0 [125.0 to 282.0] | 146.5 [82.5 to 223.5]
  Week 40, n=50, 48, 47, 44: number analyzed (Participants) | 50 | 48 | 47 | 44
  Week 40, n=50, 48, 47, 44 | 205.0 [136.0 to 364.0] | 204.5 [157.5 to 346.5] | 224.0 [123.0 to 322.0] | 171.5 [123.0 to 268.0]
  Week 48, n=51, 47, 47, 45: number analyzed (Participants) | 51 | 47 | 47 | 45
  Week 48, n=51, 47, 47, 45 | 204.0 [127.0 to 384.0] | 249.0 [143.0 to 416.0] | 223.0 [141.0 to 292.0] | 174.0 [91.0 to 292.0]
  Week 60, n=51, 48, 47, 43: number analyzed (Participants) | 51 | 48 | 47 | 43
  Week 60, n=51, 48, 47, 43 | 265.0 [173.0 to 365.0] | 278.0 [198.5 to 369.5] | 229.0 [166.0 to 306.0] | 221.0 [153.0 to 355.0]
  Week 72, n=51, 47, 48, 44: number analyzed (Participants) | 51 | 47 | 48 | 44
  Week 72, n=51, 47, 48, 44 | 236.0 [177.0 to 351.0] | 285.0 [186.0 to 427.0] | 220.0 [146.0 to 373.0] | 195.0 [144.0 to 334.5]
  Week 84, n=51, 47, 46, 42: number analyzed (Participants) | 51 | 47 | 46 | 42
  Week 84, n=51, 47, 46, 42 | 292.0 [222.0 to 408.0] | 313.0 [244.0 to 366.0] | 280.0 [197.0 to 379.0] | 296.5 [187.0 to 400.0]
  Week 96, n=48, 44, 46, 39: number analyzed (Participants) | 48 | 44 | 46 | 39
  Week 96, n=48, 44, 46, 39 | 335.0 [253.5 to 478.5] | 391.5 [243.0 to 527.0] | 326.0 [236.0 to 451.0] | 301.0 [204.0 to 445.0]

5. Secondary Outcome: Number of Participants With New HIV-associated Conditions of the Indicated Class
Description: HIV-associated conditions were assessed according to the Centers for Disease Control and Prevention (CDC) HIV-1 classification system. Category (CAT) A: one or more of the following conditions (CON), without any CON listed in Categories B and C: asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have a clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C: the clinical CON listed in the acquired immunodeficiency syndrome (AIDS) surveillance case definition.
Time Frame: From Baseline up to Week 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Participants
  Category B | 2 | 0 | 1 | 1
  Category C | 0 | 0 | 1 | 0
  Death | 1 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With the Indicated Type of HIV-1 Disease Progression (AIDS or Death)
Description: Clinical disease progression (CDP) was assessed according to the Centers for Disease Control and Prevention (CDC) HIV-1 classification system. Category (CAT) A: one or more of the following conditions (CON), without any CON listed in Categories B and C: asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have a clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C: the clinical CON listed in the AIDS surveillance case definition. Indicators of CDP were defined as: CAT A at Baseline (BS) to CAT B event (EV), CAT A at BS to a CAT C EV; CAT B at BS to a CAT C EV; CAT C at BS to a new CAT C EV; or CAT A, B, or C at BS to death.
Time Frame: From Baseline up to Week 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Participants
  CAT A at Baseline to a CAT C event | 0 | 0 | 0 | 0
  CAT B at Baseline to a CAT C event | 0 | 0 | 1 | 0
  CAT C at Baseline to a new CAT C event | 0 | 0 | 0 | 0
  CAT A, B, or C at Baseline to death | 1 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 c/mL
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1), Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, Week 84, and Week 96. The analysis was performed using the time to loss of virological response (TLOVR) dataset. In the TLOVR dataset, participant responses at a specified threshold of HIV-1 RNA (<50 copies/mL) are determined by using the Food and Drug Administration's TLOVR algorithm. Using the TLOVR algorithm, participants are considered to have failed on therapy if they never achieved confirmed RNA levels below the threshold, if they had confirmed rebound of RNA above the threshold, if they made a non-permitted change in background regimen, or if they permanently discontinued investigational product for any reason.
Time Frame: as for outcome 3
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Participants
  Baseline | 0 | 0 | 0 | 0
  Week 1 | 6 | 4 | 4 | 3
  Week 2 | 22 | 19 | 11 | 6
  Week 4 | 37 | 35 | 31 | 9
  Week 8 | 46 | 45 | 43 | 18
  Week 12 | 50 | 46 | 45 | 25
  Week 16 | 51 | 46 | 47 | 29
  Week 20 | 51 | 47 | 47 | 38
  Week 24 | 51 | 46 | 47 | 41
  Week 32 | 50 | 45 | 46 | 43
  Week 40 | 49 | 45 | 46 | 42
  Week 48 | 48 | 45 | 46 | 40
  Week 60 | 48 | 44 | 46 | 41
  Week 72 | 48 | 44 | 45 | 40
  Week 84 | 47 | 43 | 46 | 38
  Week 96 | 42 | 40 | 45 | 36

8. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <400 c/mL
Description: Plasma samples were collected for quantitative HIV-1 RNA analysis at Baseline (Day 1), Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, Week 84, and Week 96. The analysis was performed using the time to loss of virological response (TLOVR) dataset. In the TLOVR dataset, participant responses at a specified threshold of HIV-1 RNA (<400 c/mL) are determined by using the Food and Drug Administration's TLOVR algorithm. Using the TLOVR algorithm, participants are considered to have failed on therapy if they never achieved confirmed RNA levels below the threshold, if they had confirmed rebound of RNA above the threshold, if they made a non-permitted change in background regimen, or if they permanently discontinued investigational product for any reason.
Time Frame: as for outcome 3
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Participants
  Baseline | 0 | 0 | 0 | 0
  Week 1 | 25 | 20 | 16 | 15
  Week 2 | 45 | 45 | 41 | 23
  Week 4 | 52 | 49 | 48 | 32
  Week 8 | 52 | 49 | 49 | 41
  Week 12 | 52 | 49 | 49 | 45
  Week 16 | 52 | 48 | 49 | 45
  Week 20 | 52 | 48 | 49 | 45
  Week 24 | 52 | 47 | 48 | 45
  Week 32 | 52 | 47 | 48 | 45
  Week 40 | 50 | 47 | 48 | 45
  Week 48 | 50 | 47 | 48 | 44
  Week 60 | 50 | 46 | 48 | 44
  Week 72 | 50 | 46 | 47 | 43
  Week 84 | 50 | 45 | 47 | 42
  Week 96 | 46 | 43 | 46 | 39

9. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Events (SAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity; or is a congenital anomaly/birth defect. All clinically suspected cases of hypersensitivity reaction to abacavir in participants receiving abacavir/lamivudine were reported as SAEs. Medical or scientific judgment was to have been exercised in other situations. Refer to the general AE/SAE module for a list of AEs (occuring at a frequency threshold >=3%) and SAEs.
Time Frame: From Baseline up to Week 96/Early Withdrawal
Population: Safety Population:All participants who received at least one dose of the study medication
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Participants
  Any AE | 50 | 46 | 46 | 46
  Any SAE | 5 | 5 | 7 | 7

10. Secondary Outcome: Number of Participants With the Indicated Grade 1 to Grade 4 Treatment-emergent Clinical Chemistry and Hematology Toxicities
Description: Blood samples were collected for the measurement of clinical chemistry and hematology parameters. Toxicities were graded for severity according to the Division of AIDS (DAIDS) toxicity scales as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (potentially life threatening).
Time Frame: From Baseline up to Week 96/Early Withdrawal
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 53 | 51 | 51 | 50
Participants
  Alanine amino transferase | 7 | 11 | 3 | 19
  Cholesterol | 18 | 16 | 13 | 24
  Creatinine kinase | 17 | 6 | 7 | 5
  Lipase | 11 | 13 | 11 | 9
  Triglycerides | 0 | 1 | 2 | 1
  Alkaline phosphatase | 1 | 0 | 1 | 10
  Amylase | 2 | 3 | 1 | 4
  Aspartate amino transferase | 12 | 8 | 6 | 9
  Carbon dioxide content/bicarbonate | 28 | 24 | 23 | 30
  Creatinine | 0 | 4 | 0 | 0
  Hypercalcemia | 0 | 0 | 0 | 1
  Hyperglycaemia | 16 | 15 | 17 | 17
  Hyperkalemia | 0 | 0 | 1 | 1
  Hypernatremia | 1 | 1 | 1 | 0
  Hypocalcemia | 4 | 5 | 5 | 8
  Hypoglycaemia | 3 | 3 | 5 | 4
  Hypokalemia | 4 | 1 | 3 | 3
  Hyponatremia | 6 | 12 | 7 | 13
  Low-density lipoprotein cholesterol | 14 | 15 | 11 | 20
  Magnesium | 7 | 6 | 5 | 4
  Phosphate, inorganic | 9 | 15 | 14 | 11
  Total bilirubin | 3 | 4 | 3 | 0
  Activated partial thromboplastin time | 7 | 12 | 6 | 5
  Hemoglobin | 0 | 1 | 0 | 1
  International normalized ratio | 6 | 9 | 6 | 5
  Platelet count | 1 | 4 | 1 | 1
  Prothrombin time | 7 | 8 | 7 | 4
  Total neutrophils | 9 | 7 | 6 | 10
  White blood cell count | 1 | 1 | 1 | 1

11. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Integrase (IN) Mutations Detected at the Time of Protocol-defined Virologic Failure (PDVF), as a Measure of Genotypic Resistance
Description: For participants meeting one of the criteria for PDVF, plasma samples collected at the time point of virologic failure were tested to evaluate any potential genotypic and/or phenotypic evolution of resistance. PDVF was defined as (A) Virologic Non-response: a decrease in plasma HIV-1 RNA of <1 log10 copies/mL by Week 4, with subsequent confirmation, unless plasma HIV-1 RNA is <400 copies/mL; confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 without evidence of prior suppression to <400copies/mL or (B) Virologic Rebound: confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL; confirmed plasma HIV-1 RNA levels >0.5 log10 copies/mL above the nadir value, where nadir is the lowest HIV-1 value >=400 copies/mL.On-treatment Genotypic Resistance Population: all participants in the ITT-E Population with available on-treatment genotypic data, excluding participants who were not protocol-defined virologic failures.
Time Frame: From Baseline up to Week 96/Early Withdrawal
Population: On-treatment Genotypic Resistance Population.
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 2 | 1 | 0 | 1
Participants
  A23A/V | 1 | 0 |  | 0
  S255N | 1 | 0 |  | 0

12. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Major Mutations of Other Classes Detected at the Time of Protocol-defined Virologic Failure (PDVF), as a Measure of Genotypic Resistance
Description: For participants meeting one of the criteria for PDVF, plasma samples collected at the time point of virologic failure were tested to evaluate any potential genotypic and/or phenotypic evolution of resistance. PDVF was defined as (A) Virologic Non-response: a decrease in plasma HIV-1 RNA of <1 log10 copies/mL by Week 4, with subsequent confirmation, unless plasma HIV-1 RNA is <400 copies/mL; confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 without evidence of prior suppression to <400copies/mL or (B) Virologic Rebound: confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL; confirmed plasma HIV-1 RNA levels >0.5 log10 copies/mL above the nadir value, where nadir is the lowest HIV-1 value >=400 copies/mL.
Time Frame: From Baseline up to Week 96/Early Withdrawal
Population: On-treatment Genotypic Resistance Population
Measure: Number; unit: Participants
Groups:
- DTG 10 mg QD: Participants received DTG 10 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg QD.
- DTG 25 mg QD: Participants received DTG 25 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg QD.
- DTG 50 mg QD: Participants received DTG 50 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg QD.
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 2 | 1 | 0 | 1
Participants | 1 | 0 |  | 0

13. Secondary Outcome: Number of Participants With the Indicated Fold Increase in DTG FC (Fold Change in IC50 Relative to Wild-type Virus) at the Time of PDVF, as a Measure of Post-Baseline Phenotypic Resistance
Description: The FC in IC50 (50% inhibitory concentration) for DTG relative to wild-type virus was determined for virus isolated at Baseline and at the time of PDVF. Fold increase in DTG FC at the time of PDVF was derived as the PDVF FC/Baseline FC ratio. PDVF was defined as (A) Virologic Non-response: a decrease in plasma HIV-1 RNA of <1 log10 copies/mL by Week 4, with subsequent confirmation, unless plasma HIV-1 RNA is <400 copies/mL; confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 without evidence of prior suppression to <400copies/mL or (B) Virologic Rebound: confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL; confirmed plasma HIV-1 RNA levels >0.5 log10 copies/mL above the nadir value, where nadir is the lowest HIV-1 value >=400 copies/mL.On-treatment Phenotypic Resistance Population: all participants in the ITT-E Population with available on-treatment phenotypic data
Time Frame: From Baseline up to Week 96/Early Withdrawal
Population: On-treatment Phenotypic Resistance Population
Measure: Number; unit: Participants
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 2 | 1 | 0 | 0
Participants
  <1 fold | 0 | 1 |  |
  1-<2 fold | 2 | 0 |  |
  2-<4 fold | 0 | 0 |  |
  4-<8 fold | 0 | 0 |  |
  >=8 fold | 0 | 0 |  |

14. Secondary Outcome: Plasma DTG Concentration
Description: Blood samples for the determination of plasma DTG concentration were collected from the participants randomized to receive DTG, at the following time points: pre-dose and 2-4 hours post-dose at Weeks 2, Week 12, and Week 24. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed. The Pharmacokinetic (PK) Summary Population is comprised of all participants who received DTG and underwent intensive PK sampling or limited PK sampling during the study and provided evaluable DTG PK parameters. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles).Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the PK Summary Population.
Time Frame: Week 2, Week 12, and Week 24
Population: PK Summary Population.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (µg/mL)
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 48 | 46 | 46 | 0
Micrograms per milliliter (µg/mL)
  Week 2, Pre-dose, n=46, 44, 43, 0: number analyzed (Participants) | 46 | 44 | 43 | 0
  Week 2, Pre-dose, n=46, 44, 43, 0 | 0.3580 (0.18321) | 0.6779 (0.44085) | 1.4044 (0.88041) |
  Week 2, 2-4 hours post-dose, n=31, 29, 29, 0: number analyzed (Participants) | 31 | 29 | 29 | 0
  Week 2, 2-4 hours post-dose, n=31, 29, 29, 0 | 1.0121 (0.28125) | 1.9716 (0.71890) | 3.8414 (1.87405) |
  Week 12, Pre-dose, n= 46, 45, 44, 0: number analyzed (Participants) | 46 | 45 | 44 | 0
  Week 12, Pre-dose, n= 46, 45, 44, 0 | 0.3648 (0.16791) | 0.5759 (0.32645) | 1.4169 (1.00152) |
  Week 12, 2-4 hours post-dose, n=48, 45, 45, 0: number analyzed (Participants) | 48 | 45 | 45 | 0
  Week 12, 2-4 hours post-dose, n=48, 45, 45, 0 | 1.0374 (0.27517) | 1.7907 (0.70953) | 3.6056 (1.33862) |
  Week 24, Pre-dose, n=45, 44, 44, 0: number analyzed (Participants) | 45 | 44 | 44 | 0
  Week 24, Pre-dose, n=45, 44, 44, 0 | 0.3766 (0.23399) | 0.6636 (0.50767) | 1.4534 (0.94283) |
  Week 24, 2-4 hours post-dose, n=45, 45, 45, 0: number analyzed (Participants) | 45 | 45 | 45 | 0
  Week 24, 2-4 hours post-dose, n=45, 45, 45, 0 | 1.0113 (0.34083) | 1.9021 (0.79430) | 3.5397 (1.36538) |

15. Secondary Outcome: AUC(0-tau) of DTG
Description: The area under the time concentration curve over the dosing interval (AUC[0-tau]) of DTG was determined using non-compartmental analysis based on intensive PK sampling at the following time points: pre-dose; 2, 3, 4, 8, and 24 hours post-dose at Week 2. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed. Only those participants available at the specified time points were analyzed.
Time Frame: Pre-dose and 2, 3, 4, 8, and 24 hours post-dose at Week 2
Population: PK Summary Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*µg/mL
Groups:
- DTG 10 mg QD: Participants received DTG 10 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg OD.
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 15 | 15 | 15 | 0
Hours*µg/mL | 16.0 (40) | 23.1 (48) | 48.1 (40) |

16. Secondary Outcome: Maximal Concentration (Cmax), Minimal Concentration (Cmin), and Concentration at the End of Dosing Interval (Ctau) of DTG
Description: The Cmax, Cmax, and Ctau of DTG were determined using non-compartmental analysis based on intensive PK sampling at the following time points: pre-dose; 2, 3, 4, 8, and 24 hours post-dose at Week 2. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed.
Time Frame: Pre-dose and 2, 3, 4, 8, and 24 hours post-dose at Week 2
Population: PK Summary Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- DTG 10 mg OD: Participants received DTG 10 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally OD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg OD.
- DTG 25 mg OD: Participants received DTG 25 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally OD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg OD.
- DTG 50 mg OD: Participants received DTG 50 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally OD for 96 weeks. Following Week 96, participants continued to receive DTG 50 mg OD.
- EFV 600 mg OD: Participants received Efavirenz (EFV) 600 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally OD for 96 weeks.
Arm/Group | DTG 10 mg OD | DTG 25 mg OD | DTG 50 mg OD | EFV 600 mg OD
Number analyzed (Participants) | 15 | 15 | 15 | 0
µg/mL
  Cmax | 1.10 (37) | 1.71 (43) | 3.40 (27) |
  Cmin | 0.33 (64) | 0.44 (68) | 0.94 (74) |
  Ctau | 0.37 (55) | 0.45 (71) | 1.05 (72) |

17. Secondary Outcome: Pre-dose Concentration (C0) and C0 Avg of DTG
Description: The plasma DTG C0 of DTG was determined using limited/sparse PK sampling at Week 2, Week 12, and Week 24. C0 avg was calculated at Week 24 as the mean of the C0 of DTG at Week 2, Week 12, and Week 24. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the PK Summary Population.
Time Frame: Week 2, Week 12, and Week 24
Population: PK Summary Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (µg/mL)
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 49 | 46 | 46 | 0
Microgram per milliliter (µg/mL)
  C0, Week 2, n=46, 44, 43, 0: number analyzed (Participants) | 46 | 44 | 43 | 0
  C0, Week 2, n=46, 44, 43, 0 | 0.31 (58) | 0.57 (62) | 1.20 (61) |
  C0, Week 12, n=46, 45, 44, 0: number analyzed (Participants) | 46 | 45 | 44 | 0
  C0, Week 12, n=46, 45, 44, 0 | 0.33 (49) | 0.47 (77) | 1.13 (95) |
  C0, Week 24, n=45, 44, 44, 0: number analyzed (Participants) | 45 | 44 | 44 | 0
  C0, Week 24, n=45, 44, 44, 0 | 0.33 (67) | 0.57 (74) | 1.20 (74) |
  C0 avg, n=48, 46, 46, 0: number analyzed (Participants) | 48 | 46 | 46 | 0
  C0 avg, n=48, 46, 46, 0 | 0.34 (49) | 0.56 (61) | 1.25 (55) |

18. Secondary Outcome: Time to Maximal Drug Concentration (Tmax) of DTG
Description: Tmax of DTG was determined using non-compartmental analysis based on intensive PK sampling at the following time points: pre-dose; 2, 3, 4, 8, and 24 hours post-dose at Week 2. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed.
Time Frame: Pre-dose and 2, 3, 4, 8, and 24 hours post-dose at Week 2
Population: PK Summary Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 15 | 15 | 15 | 0
Hours | 2.0 [2.0 to 4.0] | 2.0 [2.0 to 8.0] | 2.0 [1.9 to 4.0] |

19. Secondary Outcome: Relationship Between the Change From Baseline in Plasma HIV-1 RNA at Week 2 and the Indicated Plasma DTG PK Parameters
Description: Relationships between Week 2 plasma DTG PK parameters (AUC[0-tau] [area under the time concentration curve over the dosing interval], Cmax [maximal concentration], and Ctau [concentration at the end of the dosing interval]) and the change from Baseline in plasma HIV-1 RNA at Week 2 (calculated as the post-Baseline value minus the value at Baseline) was assessed using Pearson's correlation analyses. The Pearson's correlation coefficient is a measure of the correlation between plasma HIV-1 RNA and plasma DTG PK parameters and ranges from -1 to 1. A value of 0 indicates no statistical association; a value close to -1 or 1 indicates a higher association. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed. PK/Pharmacodynamic (PD) Analysis Population: all participants with available PD measures (e.g., safety and/or efficacy data) and with evaluable DTG plasma concentration data considered suitable for investigation of relationship with the PD measures
Time Frame: Week 2
Population: PK/PD Analysis Population.Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Pearson's correlation coefficient
Groups:
- Overall DTG: All participants who received DTG in any DTG treatment group (DTG 10 mg QD, DTG 25 mg QD, and DTG 50 mg QD)
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD | Overall DTG
Number analyzed (Participants) | 15 | 15 | 15 | 0 | 45
Pearson's correlation coefficient
  AUC(0-tau) | 0.426 | -0.018 | -0.258 |  | -0.086
  Cmax | 0.452 | -0.051 | -0.150 |  | -0.055
  Ctau | 0.273 | -0.100 | -0.263 |  | -0.129

20. Secondary Outcome: Relationship Between the Change From Baseline in CD4+ Cell Counts at Week 96 and the Indicated Plasma DTG PK Parameters
Description: Relationships between plasma DTG PK parameters (AUC[0-tau] [area under the time concentration curve over the dosing interval], Cmax [maximal concentration], C0avg [average pre-dose concentration], and Ctau [concentration at the end of the dosing interval]) and the change from Baseline in CD4+ cell counts at Week 96 (calculated as the post-Baseline value minus the value at Baseline) was assessed using Pearson's correlation analyses. The Pearson's correlation coefficient is a measure of the correlation between CD4+ cell counts and plasma DTG PK parameters and ranges from -1 to 1. A value of 0 indicates no statistical association; a value close to -1 or 1 indicates a higher association.Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed.Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Time Frame: Week 96
Population: PK/PD Analysis Population.
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD | Overall DTG
Number analyzed (Participants) | 50 | 46 | 46 | 0 | 142
Pearson's correlation coefficient
  AUC(0-tau), n=13, 14, 15, 0: number analyzed (Participants) | 13 | 14 | 15 | 0 | 142
  AUC(0-tau), n=13, 14, 15, 0 | -0.100 | 0.379 | 0.008 |  | -0.005
  Cmax, n=13, 14, 15, 0: number analyzed (Participants) | 13 | 14 | 15 | 0 | 142
  Cmax, n=13, 14, 15, 0 | -0.047 | 0.332 | 0.234 |  | 0.037
  C0avg, n=43, 40, 42, 0: number analyzed (Participants) | 43 | 40 | 42 | 0 | 142
  C0avg, n=43, 40, 42, 0 | -0.009 | -0.013 | 0.206 |  | -0.011
  Ctau, n=13, 14, 15, 0: number analyzed (Participants) | 13 | 14 | 15 | 0 | 142
  Ctau, n=13, 14, 15, 0 | -0.289 | 0.299 | -0.074 |  | -0.055

21. Secondary Outcome: Relationship Between the Indicated Safety Parameters at Week 96 and the Indicated Plasma DTG PK Parameters
Description: Relationships between log-transformed plasma DTG PK parameters (AUC[0-tau], Cmax, C0, C0avg, Ctau, and Cmin) and safety parameters (AE occurrence, maximum AE intensity, alanine aminotransferase [ALT], change from Baseline [CFB] in ALT, total bilirubin, CFB in total bilirubin, creatine kinase, CFB in creatine kinase, triglycerides, CFB in triglycerides, lipase, CFB in lipase, total cholesterol [TC], CFB in TC) was assessed using Pearson's correlation analyses. The Pearson's correlation coefficient is a measure of the correlation between safety parameters and plasma DTG PK parameters and ranges from -1 to 1. A value of 0 indicates no statistical association; a value close to -1 or 1 indicates a higher association. The presence of >=1 AE was used for AE occurrence. The most severe AE grade/intensity was used for maximum AE intensity. Maximum laboratory values per participant were used for safety parameters. CFB was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Week 96
Population: PK/PD Analysis Population.Only those participants available at the specified time points were analyzed
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | Overall DTG
Number analyzed (Participants) | 142
Pearson's correlation coefficient
  AUC(0-tau) versus AE occurrence, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus AE occurrence, n=45 | 0.114
  AUC(0-tau) versus maximum AE intensity, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus maximum AE intensity, n=45 | 0.171
  AUC(0-tau) versus ALT, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus ALT, n=45 | -0.196
  AUC(0-tau) versus CFB in ALT, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus CFB in ALT, n=45 | -0.201
  AUC(0-tau) versus total bilirubin, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus total bilirubin, n=45 | 0.364
  AUC(0-tau) versus CFB in total bilirubin, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus CFB in total bilirubin, n=45 | 0.147
  AUC(0-tau) versus creatine kinase, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus creatine kinase, n=45 | -0.168
  AUC(0-tau) versus CFB in creatine kinase, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus CFB in creatine kinase, n=45 | -0.145
  AUC(0-tau) vs Triglycerides, n=45: number analyzed (Participants) | 45
  AUC(0-tau) vs Triglycerides, n=45 | 0.104
  AUC(0-tau) versus CFB in triglycerides, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus CFB in triglycerides, n=45 | 0.216
  AUC(0-tau) versus lipase, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus lipase, n=45 | -0.066
  AUC(0-tau) versus CFB in lipase, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus CFB in lipase, n=45 | 0.092
  AUC(0-tau) versus total cholesterol, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus total cholesterol, n=45 | -0.097
  AUC(0-tau) versus CFB in total cholesterol, n=45: number analyzed (Participants) | 45
  AUC(0-tau) versus CFB in total cholesterol, n=45 | -0.153
  Cmax versus AE occurrence, n=45: number analyzed (Participants) | 45
  Cmax versus AE occurrence, n=45 | 0.061
  Cmax versus maximum AE intensity, n=45: number analyzed (Participants) | 45
  Cmax versus maximum AE intensity, n=45 | 0.110
  Cmax versus ALT, n=45: number analyzed (Participants) | 45
  Cmax versus ALT, n=45 | -0.135
  Cmax versus CFB in ALT, n=45: number analyzed (Participants) | 45
  Cmax versus CFB in ALT, n=45 | -0.135
  Cmax versus total bilirubin, n=45: number analyzed (Participants) | 45
  Cmax versus total bilirubin, n=45 | 0.265
  Cmax versus CFB in total bilirubin, n=45: number analyzed (Participants) | 45
  Cmax versus CFB in total bilirubin, n=45 | 0.033
  Cmax versus creatine kinase, n=45: number analyzed (Participants) | 45
  Cmax versus creatine kinase, n=45 | -0.188
  Cmax versus CFB in creatine kinase, n=45: number analyzed (Participants) | 45
  Cmax versus CFB in creatine kinase, n=45 | -0.161
  Cmax versus triglycerides, n=45: number analyzed (Participants) | 45
  Cmax versus triglycerides, n=45 | 0.134
  Cmax versus CFB in triglycerides, n=45: number analyzed (Participants) | 45
  Cmax versus CFB in triglycerides, n=45 | 0.244
  Cmax versus lipase, n=45: number analyzed (Participants) | 45
  Cmax versus lipase, n=45 | -0.034
  Cmax versus CFB in lipase, n=45: number analyzed (Participants) | 45
  Cmax versus CFB in lipase, n=45 | 0.115
  Cmax versus total cholesterol, n=45: number analyzed (Participants) | 45
  Cmax versus total cholesterol, n=45 | -0.101
  Cmax versus CFB in total cholesterol, n=45: number analyzed (Participants) | 45
  Cmax versus CFB in total cholesterol, n=45 | -0.192
  C0 versus AE occurrence, n=133: number analyzed (Participants) | 133
  C0 versus AE occurrence, n=133 | -0.080
  C0 versus maximum AE intensity, n=133: number analyzed (Participants) | 133
  C0 versus maximum AE intensity, n=133 | -0.003
  C0 versus ALT, n=133: number analyzed (Participants) | 133
  C0 versus ALT, n=133 | -0.196
  C0 versus CFB in ALT, n=133: number analyzed (Participants) | 133
  C0 versus CFB in ALT, n=133 | -0.237
  C0 versus total bilirubin, n=133: number analyzed (Participants) | 133
  C0 versus total bilirubin, n=133 | 0.298
  C0 versus CFB in total bilirubin, n=133: number analyzed (Participants) | 133
  C0 versus CFB in total bilirubin, n=133 | 0.120
  C0 versus creatine kinase, n=133: number analyzed (Participants) | 133
  C0 versus creatine kinase, n=133 | -0.094
  C0 versus CFB in creatine kinase, n=133: number analyzed (Participants) | 133
  C0 versus CFB in creatine kinase, n=133 | -0.093
  C0 versus triglycerides, n=133: number analyzed (Participants) | 133
  C0 versus triglycerides, n=133 | -0.058
  C0 versus CFB in triglycerides, n=133: number analyzed (Participants) | 133
  C0 versus CFB in triglycerides, n=133 | -0.012
  C0 versus lipase, n=133: number analyzed (Participants) | 133
  C0 versus lipase, n=133 | -0.187
  C0 versus CFB in lipase, n=133: number analyzed (Participants) | 133
  C0 versus CFB in lipase, n=133 | -0.137
  C0 versus total cholesterol, n=133: number analyzed (Participants) | 133
  C0 versus total cholesterol, n=133 | -0.179
  C0 versus CFB in total cholesterol, n=133: number analyzed (Participants) | 133
  C0 versus CFB in total cholesterol, n=133 | -0.125
  C0avg versus AE occurrence, n=140: number analyzed (Participants) | 140
  C0avg versus AE occurrence, n=140 | -0.028
  C0avg versus maximum AE intensity, n=140: number analyzed (Participants) | 140
  C0avg versus maximum AE intensity, n=140 | 0.036
  C0avg versus ALT, n=140: number analyzed (Participants) | 140
  C0avg versus ALT, n=140 | -0.166
  C0avg versus CFB in ALT, n=140: number analyzed (Participants) | 140
  C0avg versus CFB in ALT, n=140 | -0.177
  C0avg versus total bilirubin, n=140: number analyzed (Participants) | 140
  C0avg versus total bilirubin, n=140 | 0.319
  C0avg versus CFB in total bilirubin, n=140: number analyzed (Participants) | 140
  C0avg versus CFB in total bilirubin, n=140 | 0.109
  C0avg versus creatine kinase, n=140: number analyzed (Participants) | 140
  C0avg versus creatine kinase, n=140 | -0.114
  C0avg versus CFB in creatine kinase, n=140: number analyzed (Participants) | 140
  C0avg versus CFB in creatine kinase, n=140 | -0.110
  C0avg versus triglycerides, n=140: number analyzed (Participants) | 140
  C0avg versus triglycerides, n=140 | 0.057
  C0avg versus CFB in triglycerides, n=140: number analyzed (Participants) | 140
  C0avg versus CFB in triglycerides, n=140 | 0.092
  C0avg versus lipase, n=140: number analyzed (Participants) | 140
  C0avg versus lipase, n=140 | -0.164
  C0avg versus CFB in lipase, n=140: number analyzed (Participants) | 140
  C0avg versus CFB in lipase, n=140 | -0.120
  C0avg versus total cholesterol, n=140: number analyzed (Participants) | 140
  C0avg versus total cholesterol, n=140 | -0.170
  C0avg versus CFB in total cholesterol, n=140: number analyzed (Participants) | 140
  C0avg versus CFB in total cholesterol, n=140 | -0.083
  Ctau versus AE occurrence, n=45: number analyzed (Participants) | 45
  Ctau versus AE occurrence, n=45 | 0.190
  Ctau versus maximum AE intensity, n=45: number analyzed (Participants) | 45
  Ctau versus maximum AE intensity, n=45 | 0.205
  Ctau versus ALT, n=45: number analyzed (Participants) | 45
  Ctau versus ALT, n=45 | -0.281
  Ctau versus CFB in ALT, n=45: number analyzed (Participants) | 45
  Ctau versus CFB in ALT, n=45 | -0.285
  Ctau versus total bilirubin, n=45: number analyzed (Participants) | 45
  Ctau versus total bilirubin, n=45 | 0.446
  Ctau versus CFB in total bilirubin, n=45: number analyzed (Participants) | 45
  Ctau versus CFB in total bilirubin, n=45 | 0.237
  Ctau versus creatine kinase, n=45: number analyzed (Participants) | 45
  Ctau versus creatine kinase, n=45 | -0.143
  Ctau versus CFB in creatine kinase, n=45: number analyzed (Participants) | 45
  Ctau versus CFB in creatine kinase, n=45 | -0.125
  Ctau versus triglycerides, n=45: number analyzed (Participants) | 45
  Ctau versus triglycerides, n=45 | 0.061
  Ctau versus CFB in triglycerides, n=45: number analyzed (Participants) | 45
  Ctau versus CFB in triglycerides, n=45 | 0.172
  Ctau versus lipase, n=45: number analyzed (Participants) | 45
  Ctau versus lipase, n=45 | -0.131
  Ctau versus CFB in lipase, n=45: number analyzed (Participants) | 45
  Ctau versus CFB in lipase, n=45 | 0.056
  Ctau versus total cholesterol, n=45: number analyzed (Participants) | 45
  Ctau versus total cholesterol, n=45 | -0.039
  Ctau versus CFB in total cholesterol, n=45: number analyzed (Participants) | 45
  Ctau versus CFB in total cholesterol, n=45 | -0.108
  Cmin versus AE occurrence, n=45: number analyzed (Participants) | 45
  Cmin versus AE occurrence, n=45 | 0.156
  Cmin versus maximum AE intensity, n=45: number analyzed (Participants) | 45
  Cmin versus maximum AE intensity, n=45 | 0.193
  Cmin versus ALT, n=45: number analyzed (Participants) | 45
  Cmin versus ALT, n=45 | -0.236
  Cmin versus CFB in ALT, n=45: number analyzed (Participants) | 45
  Cmin versus CFB in ALT, n=45 | -0.253
  Cmin versus total bilirubin, n=45: number analyzed (Participants) | 45
  Cmin versus total bilirubin, n=45 | 0.430
  Cmin versus CFB in total bilirubin, n=45: number analyzed (Participants) | 45
  Cmin versus CFB in total bilirubin, n=45 | 0.171
  Cmin versus creatine kinase, n=45: number analyzed (Participants) | 45
  Cmin versus creatine kinase, n=45 | -0.132
  Cmin versus CFB in creatine kinase, n=45: number analyzed (Participants) | 45
  Cmin versus CFB in creatine kinase, n=45 | -0.124
  Cmin versus triglycerides, n=45: number analyzed (Participants) | 45
  Cmin versus triglycerides, n=45 | -0.042
  Cmin versus CFB in triglycerides, n=45: number analyzed (Participants) | 45
  Cmin versus CFB in triglycerides, n=45 | 0.057
  Cmin versus lipase, n=45: number analyzed (Participants) | 45
  Cmin versus lipase, n=45 | -0.135
  Cmin versus CFB in lipase, n=45: number analyzed (Participants) | 45
  Cmin versus CFB in lipase, n=45 | 0.032
  Cmin versus total cholesterol, n=45: number analyzed (Participants) | 45
  Cmin versus total cholesterol, n=45 | -0.194
  Cmin versus CFB in total cholesterol, n=45: number analyzed (Participants) | 45
  Cmin versus CFB in total cholesterol, n=45 | -0.208

22. Secondary Outcome: Relationship Between Gastrointestinal System Organ Class AEs of Special Interest at Week 96 and the Indicated Plasma DTG PK Parameters
Description: Logistic regressions were performed to examine the correlation between plasma DTG PK parameters (AUC[0-tau] [area under the time concentration curve over the dosing interval], Cmax [maximal concentration], Ctau [concentration at the end of the dosing interval], and C0avg [average pre-dose concentration]) on log scales and the presence of gastrointestinal system organ class AEs (abdominal pain, diarrhea, nausea, and vomiting) at Week 96. Data are presented as estimates from logistic regression, which is a measure of the association between AEs of special interest and plasma DTG PK parameters. A value of 0 indicates no statistical association; a large absolute value of the estimate indicates higher association. Because PK was assessed for DTG, no participants in the EFV treatment group were analyzed. Results are presented for participants in any DTG group (overall DTG).Only those participants available at the specified time points were analyzed represented by n=X in the category titles
Time Frame: Week 96
Population: PK/PD Analysis Population.
Measure: Number; unit: estimated effect
Groups:
- Overall DTG: All participants who received DTG in any DTG treatment group (DTG 10 mg OD, DTG 25 mg OD, and DTG 50 mg OD).
Arm/Group | Overall DTG
Number analyzed (Participants) | 142
estimated effect
  Abdominal pain versus AUC(0-tau), n=45: number analyzed (Participants) | 45
  Abdominal pain versus AUC(0-tau), n=45 | -2.49
  Abdominal pain versus Cmax, n=45: number analyzed (Participants) | 45
  Abdominal pain versus Cmax, n=45 | -2.98
  Abdominal pain versus Ctau, n=45: number analyzed (Participants) | 45
  Abdominal pain versus Ctau, n=45 | -1.72
  Abdominal pain versus C0avg, n=140: number analyzed (Participants) | 140
  Abdominal pain versus C0avg, n=140 | -0.41
  Diarrhoea versus AUC(0-tau), n=45: number analyzed (Participants) | 45
  Diarrhoea versus AUC(0-tau), n=45 | -0.62
  Diarrhoea versus Cmax, n=45: number analyzed (Participants) | 45
  Diarrhoea versus Cmax, n=45 | -0.98
  Diarrhoea versus Ctau, n=45: number analyzed (Participants) | 45
  Diarrhoea versus Ctau, n=45 | -0.29
  Diarrhoea versus C0avg, n=140: number analyzed (Participants) | 140
  Diarrhoea versus C0avg, n=140 | 0.13
  Nausea versus AUC(0-tau), n=45: number analyzed (Participants) | 45
  Nausea versus AUC(0-tau), n=45 | -0.31
  Nausea versus Cmax, n=45: number analyzed (Participants) | 45
  Nausea versus Cmax, n=45 | -0.72
  Nausea versus Ctau, n=45: number analyzed (Participants) | 45
  Nausea versus Ctau, n=45 | 0.03
  Nausea versus C0avg, n=140: number analyzed (Participants) | 140
  Nausea versus C0avg, n=140 | -0.32
  Vomiting versus AUC(0-tau), n=45: number analyzed (Participants) | 45
  Vomiting versus AUC(0-tau), n=45 | -1.29
  Vomiting versus Cmax, n=45: number analyzed (Participants) | 45
  Vomiting versus Cmax, n=45 | -1.61
  Vomiting versus Ctau, n=45: number analyzed (Participants) | 45
  Vomiting versus Ctau, n=45 | -1.15
  Vomiting versus C0avg, n=140: number analyzed (Participants) | 140
  Vomiting versus C0avg, n=140 | -0.89

23. Other Pre Specified Outcome: Change From Baseline in Cluster of Differentiation 8+ (CD8+) Cell Counts at the Indicated Time Points
Description: Change from Baseline in CD8+ cell count data are not available; CD8+ data are only listed on a per-participant basis and were not summarized.
Time Frame: as for outcome 3
Population: ITT-E Population
Arm/Group | DTG 10 mg QD | DTG 25 mg QD | DTG 50 mg QD | EFV 600 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected in the time period from Baseline up to end of study.
Description: SAEs and AEs were collected in members of Safety Population, comprised of all participants who received at least one dose of study medication.
Groups:
- DTG 10mg QD: Participants received DTG 10 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- DTG 25mg QD: Participants received DTG 25 mg, DTG matching placebo, and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- DTG 50mg QD: Participants received DTG 50 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
- EFV 600mg: Participants received Efavirenz (EFV) 600 mg and ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg orally QD for 96 weeks.
Arm/Group | DTG 10mg QD | DTG 25mg QD | DTG 50mg QD | EFV 600mg | Open-label DTG 50 mg QD
All-Cause Mortality (participants affected / at risk) | 2/53 | 0/51 | 0/51 | 0/50 | 2/138
Serious Adverse Events (participants affected / at risk) | 6/53 | 4/51 | 7/51 | 7/50 | 16/138
Other Adverse Events (participants affected / at risk) | 49/53 | 46/51 | 45/51 | 46/50 | 112/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 10mg QD (N=53) | DTG 25mg QD (N=51) | DTG 50mg QD (N=51) | EFV 600mg (N=50) | Open-label DTG 50 mg QD (N=138)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipomatosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 10mg QD (N=53) | DTG 25mg QD (N=51) | DTG 50mg QD (N=51) | EFV 600mg (N=50) | Open-label DTG 50 mg QD (N=138)
Viral upper respiratory tract infection (Infections and infestations) | 7 (10) | 7 (10) | 6 (10) | 5 (7) | 20 (27)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (10) | 7 (8) | 5 (7) | 12 (14)
Nausea (Gastrointestinal disorders) | 10 (10) | 8 (9) | 6 (6) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 7 (9) | 6 (10) | 8 (12) | 3 (5) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 6 (8) | 2 (2) | 10 (12)
Bronchitis (Infections and infestations) | 5 (7) | 2 (3) | 2 (3) | 5 (6) | 10 (14)
Insomnia (Psychiatric disorders) | 0 (0) | 7 (7) | 6 (6) | 6 (6) | 5 (5)
Influenza (Infections and infestations) | 5 (5) | 5 (6) | 4 (4) | 3 (3) | 6 (9)
Depression (Psychiatric disorders) | 3 (3) | 6 (6) | 2 (3) | 5 (5) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 2 (2) | 4 (5) | 10 (10)
Dizziness (Nervous system disorders) | 2 (2) | 3 (4) | 3 (3) | 11 (13) | 2 (2)
Syphilis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 12 (15)
Pyrexia (General disorders) | 5 (5) | 4 (4) | 1 (1) | 4 (5) | 6 (9)
Respiratory tract infection (Infections and infestations) | 4 (6) | 1 (2) | 2 (3) | 3 (4) | 9 (13)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4) | 6 (8) | 1 (1) | 7 (10)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3) | 2 (2) | 6 (6) | 2 (2)
Fatigue (General disorders) | 2 (2) | 4 (7) | 2 (2) | 6 (6) | 3 (4)
Sinusitis (Infections and infestations) | 2 (3) | 2 (3) | 3 (4) | 4 (6) | 6 (6)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (2) | 2 (2) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 5 (5)
Pharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Asthenia (General disorders) | 4 (4) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (7)
Tonsillitis (Infections and infestations) | 3 (10) | 1 (1) | 0 (0) | 1 (2) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 3 (4) | 1 (4) | 0 (0) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (5)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Gonorrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypogonadism (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Loss of libido (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Papilloma viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shigella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal pap smear abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal sphincter hypertonia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle impingement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial fibrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bulimia nervosa (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fat redistribution (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling drunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphogranuloma venereum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic atrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peyronie's disease (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presbyacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Primary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rubella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Substance use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue biting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxocariasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethritis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary sediment present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.